CLINICAL TRIAL: NCT06772831
Title: Cognitive Reappraisal Training Targeting Emotion Circuits As a Therapeutic Intervention in Borderline Patients
Brief Title: Cognitive Reappraisal Training for Borderline Personality (BPD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: William Marsh Rice University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Harold W Koenigsberg, MD, Professor of Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-0432-00001-03; 4R33MH125130-03 (NIH)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Borderline Personality Disorder
Keywords: BPD; Treatment; fMRI; Cognitive Reappraisal; Emotion Regulation; Borderline Personality
MeSH Terms: conditions — Borderline Personality Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: In the proposed study, the researchers will compare the effect of cognitive reappraisal training to a control condition in activating brain regions implicated in emotion regulation and in downregulating negative emotions. The researchers will further develop the treatment manual with BPD patients - treatment delivered 2 times a week for 6-weeks. All subjects will be seen for 6 weeks with the full battery of assessments, including fMRI imaging, carried out at baseline and the 6 week time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Reappraisal-by-Distancing (CRD) (Experimental): Patients will be coached to use cognitive reappraisal-by-distancing to downregulate their negative reactions to aversive emotional pictures using practice pictures.
  Interventions: Behavioral: Cognitive Reappraisal by Distancing
- Downregulate Condition (CD) (Active Comparator): Patients will be coached to practice their customary emotion regulatory techniques in a treatment occurring twice a week for 6 weeks.
  Interventions: Behavioral: Downregulate condition

INTERVENTIONS:
Behavioral: Cognitive Reappraisal by Distancing — Reappraisal-by-distancing treatment. Patients meet 2 times a week for 6 weeks to learn reappraisal by distancing through repeated practice with negative emotional pictures. The therapist will help model and shape the technique.
  Arms: Cognitive Reappraisal-by-Distancing (CRD)
Behavioral: Downregulate condition — Patients either meet 2x a week for 6- weeks to gain added practice, under the guidance of a therapist, using their customary emotion regulatory strategies to downregulate their negative reactions to aversive pictures.
  Arms: Downregulate Condition (CD)

SUMMARY:
Previous work by the group convinced the researchers to pursue development of focused cognitive reappraisal training as a novel approach to treatment of BPD, either as stand-alone treatment or in concert with evidence-based treatments of BPD. The present proposal aims to refine and test a proposed clinical intervention for BPD patients, training in reappraisal-by-distancing, in terms of its ability to influence hypothesized neural and behavioral targets and, once that is established, to demonstrate its ability improve clinically relevant outcome measures.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a prevalent, enduring and disabling psychiatric condition found in approximately 2% to 5.9% of the population and 20% of hospitalized psychiatric patients. Suicide rates of approximately 10% have been reported. One of the most prominent clinical features of BPD is extreme mood shifts occurring in response to external social/emotional events. The emotional instability in BPD contributes to many of the most disabling, even life-threatening, symptoms of the disorder, including suicidality, outbursts of intense anger, and seriously impaired role functioning. The severity of the BPD symptom profile, its prevalence, chronicity and high burden upon health care services make the development of effective and accessible treatment for BPD a high priority. Yet there is no current medication treatment indicated for BPD and the psychotherapies recognized for the disorder have been shown to have small effect sizes and are of limited availability. The present study builds upon work by the group that has shown that deficiencies in the ability to regulate emotion by engaging typically adaptive cognitive strategies (cognitive reappraisal, CR) and to effectively activate associated neural systems can be corrected by focused training in CR. The R61 phase of this study examines a manualized intensive training program in CR, tests that it effects target neural systems implicated in emotional processing and enhances behavioral reappraisal success. It examines 2-, 4- and 6- weeks of twice a week treatment to identify the optimal dose. Measures include fMRI imaging and clinical ratings at baseline and each of these subsequent time points. Upon demonstrating that CR training is superior to a control condition in enhancing performance in the neural target at one or more of these dose durations, the researchers will proceed to the R33 phase. In the R33 phase, the researchers will treat a larger sample of BPD patients at the optimal 6-week dose defined in the R61 phase to 1) demonstrate reproducibility of the R61 findings, 2) to demonstrate that CR training is superior to control in improving BPD clinical outcomes at the end of treatment and at 1- and 4- month follow-up, and 3) that change in activity at the neural targets is associated with clinical improvement. The results of this study can support the introduction of CR training as a new psychosocial approach for the treatment of BPD, either as stand-alone treatment or as an augmenting strategy. It may, moreover, have application to a range of psychiatric disorders characterized by severe emotional instability.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy men and women with Borderline Personality Disorder who are mentally competent and give informed voluntary written consent.
* Participants will be between the ages of 18 and 55.
* Within these requirements, the inclusion and exclusion criteria do not reflect participation based on gender or racial/ethnic group. The targeted/planned enrollment is a reflection of previous recruitment of female and ethnic minorities in other studies conducted by the PI and their colleagues and includes representations of both genders and all minorities.
* Participants with comorbid avoidant personality disorder will be included.
* Participants who meet criteria for PTSD will be included as long as they are not actively experiencing symptoms.

Exclusion Criteria:

* Participants will not meet criteria for Schizotypal Personality Disorder.
* Participants currently meeting criteria for Major Depressive Disorder will be excluded.
* BPD participants will not meet DSM-5 criteria for present PTSD, bipolar I disorder, schizophrenia, schizoaffective disorder, substance use disorder within the past 6 months, organic mental syndromes, head trauma, schizotypal personality disorder, avoidant personality disorder, CNS neurological disease, or seizure disorder. Participants meeting criteria for a non-IV substance use disorder more than 6 months prior to enrollment will not be excluded. This study allows patients who are currently taking psychotropic medications or are in psychotherapy, so long as there has been no change in medication or psychotherapy over the preceding two months.
* Participants currently meeting criteria for major depressive disorder.
* Participants meeting criteria for substance use disorder within the last 6 months or of an IV-substance use disorder at any time.
* Participants may not have a pacemaker, surgical clips, any metallic implants, or shrapnel fragments that would contraindicate MRI scanning.
* Pregnant women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Picture Induced Negative Emotion Signature (PINES) Network Activity | Baseline and 6 weeks of treatment
  Change in Picture Induced Negative Emotion Signature (PINES) network activity. by measuring neural activation using fMRI.

SECONDARY OUTCOMES:
Change in Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) Score | Baseline, 6 weeks of treatment, 1-month follow-up, and 4-month follow-up
  A validated 9-item self-report scale that assesses the severity of borderline personality disorder symptoms across four sectors: affective, cognitive, impulsive, and interpersonal. Total scores range from 0-36, with higher scores indicating greater symptom severity. Each item is rated on a 5-point scale (0-4), where 0 indicates no symptoms and 4 indicates severe symptoms.
Change in Active Lability Scale (ALS) Score | Baseline, 6 weeks of treatment, 1-month follow-up, and 4-month follow-up
  A 54-item self-report measure that assesses rapid changes in emotional states. Items are rated on a 4-point scale ranging from 0 ("very uncharacteristic of me") to 3 ("very characteristic of me"). Total scores range from 0-162, with higher scores indicating greater emotional instability.
Change in Perceived Stress Scale (PSS) | Baseline, 6 weeks of treatment, 1-month follow-up, and 4-month follow-up
  A 10-item self-report measure that assesses the degree to which situations in one's life are appraised as stressful. Items are rated on a 5-point scale from 0 ("never") to 4 ("very often"). Total scores range from 0-40, with higher scores indicating greater perceived stress.
Change in Difficulties in Emotion Regulation Scale (DERS) Scores | Baseline, 6 weeks of treatment, 1-month follow-up, and 4-month follow-up
  A 36-item self-report measure that assesses six dimensions of emotion regulation difficulties. Items are rated on a 5-point scale from 1 ("almost never") to 5 ("almost always"). Total scores range from 36-180, with higher scores indicating greater difficulties with emotion regulation.
Change in Beck Depression Inventory (BDI) Score | Baseline, 6 weeks of treatment, 1-month follow-up, and 4-month follow-up
  A 21-item self-report measure that assesses the severity of depression symptoms. Items are rated on a 4-point scale from 0-3, with total scores ranging from 0-63. Higher scores indicate more severe depressive symptoms, with scores >13 suggesting clinically significant depression.
Change in State-Trait Anxiety Inventory (STAXI) Score | Baseline, 6 weeks of treatment, 1-month follow-up, and 4-month follow-up
  A 40-item self-report measure that assesses both state anxiety (current anxiety level) and trait anxiety (general tendency to be anxious). Items are rated on a 4-point scale from 1 ("not at all") to 4 ("very much so"). Scores for each scale range from 20-80, with higher scores indicating greater anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Harold W Koenigsberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis.